CLINICAL TRIAL: NCT00705939
Title: A Multicenter, Double-Blind, Extension Trial of Two Parallel Dose Groups of Plant Cell Expressed Recombinant Human Glucocerebrosidase (prGCD) in Patients With Gaucher Disease
Brief Title: Plant Cell Expressed Recombinant Human Glucocerebrosidase Extension Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB-06-003
Expanded Access: NCT00962260 (No longer available)
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2014-07-15 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-09

CONDITIONS: Gaucher Disease
Keywords: Gaucher Disease; Enzyme replacement therapy
MeSH Terms: conditions — Gaucher Disease | interventions — taliglucerase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Naive 30 Units/kg (Experimental): Continue taliglucerase alfa treatment from PB-06-001 (NCT00376168)
  Interventions: Drug: Taliglucerase alfa
- Naive 60 Units/kg (Experimental): Continue taliglucerase alfa treatment from PB-06-001 (NCT00376168)
  Interventions: Drug: Taliglucerase alfa
- Switchover (Experimental): Continue taliglucerase alfa treatment from PB-06-002 (NCT00712348)
  Interventions: Drug: Taliglucerase alfa

INTERVENTIONS:
Drug: Taliglucerase alfa — Intravenous infusion every 2 weeks
  Other Names: Plant Cell Expressed Recombinant Human Glucocerebrosidase; prGCD

SUMMARY:
Gaucher disease, the most prevalent lysosomal storage disorder, is caused by mutations in the human glucocerebrosidase gene (GCD) leading to reduced activity of the lysosomal enzyme glucocerebrosidase and thereby to the accumulation of substrate glucocerebroside (GlcCer) in the cells of the monocyte-macrophage system.

This is an extension trial to Study NCT00376168 and NCT00712348.

DETAILED DESCRIPTION:
This will be a multi-center, double-blind, parallel group, extension trial to assess the safety and efficacy of prGCD in patients completing NCT00376168. Patients will receive IV infusion of prGCD every two weeks at the selected medical center. The duration of the extension study will be fifteen months. There will be two treatment groups: 30 units/kg every 2 weeks or 60 units/kg every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of Protocol PB-06-001
* The patient signs informed consent

Exclusion Criteria:

* Currently taking another experimental drug for any condition
* Presence of severe neurological signs and symptoms, defined as complete ocular paralysis, overt myoclonus or history of seizures, characteristic of neuronopathic Gaucher disease
* Pregnant or nursing
* Presence of any medical, emotional, behavioral or psychological condition that in the judgment of the Investigator would interfere with the patient's compliance with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-06; Primary Completion 2012-05 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (2):
  - Department of Human Genetics, Emory University School of Medicine, Decatur, Georgia
  - Neurogenetics, NYU at Rivergate, New York, New York
- Bone Marrow Transplant Service, The Royal Melbourne Hospital, Parkville, Victoria, Australia
- Mount Sinai Hospital, Toronto, Ontario, Canada
- Pontificia Universidad Catolica de Chile, Santiago, Chile
- Israel (2):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
- Morningside Medi-Clinic, Morningside, South Africa
- Hospital Universitario Miguel Servet, Zaragoza, Spain
- United Kingdom (2):
  - Lysosomal Disorders Service, Addenbrookes Hospital NHS Trust, Cambridge
  - Royal Free Hospital, London

REFERENCES:
- [Derived] Zimran A, Duran G, Mehta A, Giraldo P, Rosenbaum H, Giona F, Amato DJ, Petakov M, Munoz ET, Solorio-Meza SE, Cooper PA, Varughese S, Chertkoff R, Brill-Almon E. Long-term efficacy and safety results of taliglucerase alfa up to 36 months in adult treatment-naive patients with Gaucher disease. Am J Hematol. 2016 Jul;91(7):656-60. doi: 10.1002/ajh.24369. Epub 2016 Apr 24. PMID 27174694
- [Derived] Pastores GM, Shankar SP, Petakov M, Giraldo P, Rosenbaum H, Amato DJ, Szer J, Chertkoff R, Brill-Almon E, Zimran A. Enzyme replacement therapy with taliglucerase alfa: 36-month safety and efficacy results in adult patients with Gaucher disease previously treated with imiglucerase. Am J Hematol. 2016 Jul;91(7):661-5. doi: 10.1002/ajh.24399. Epub 2016 May 18. PMID 27102949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients completing Studies PB-06-001 (NCT00376168) or PB-06-002 (NCT00712348) were offered continued treatment in this study.
Groups:
- Naive 30 Units/kg: Patients previously naive to enzyme replacement therapy treated in Study PB-06-001 with taliglucerase alfa 30 units/kg
- Naive 60 Units/kg: Patients previously naive to enzyme replacement therapy from Study PB-06-001 treated with taliglucerase alfa 60 units/kg
- Switchover: Patients previously treated with imiglucerase in Study PB-06-002 treated with taliglucerase alfa at the same dose as their previous imiglucerase dose
Period: Overall Study
Arm/Group | Naive 30 Units/kg | Naive 60 Units/kg | Switchover
Started | 12 | 14 | 18 (1 subject enrolled but not treated in this protocol.)
Completed | 12 | 12 | 14
Not Completed | 0 | 2 | 4
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 3
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All treated patients are included in the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Naive 30 Units/kg | Naive 60 Units/kg | Switchover | Total
Number analyzed (Participants) | 12 | 14 | 18 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (11.8) | 36.6 (12.0) | 46.5 (13.7) | 41.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 9 | 22
  Male | 7 | 6 | 9 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 13 | 18 | 43
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 0 | 0 | 6 | 6
  Canada | 1 | 1 | 1 | 3
  Spain | 0 | 1 | 2 | 3
  Australia | 0 | 0 | 1 | 1
  Chile | 1 | 1 | 0 | 2
  South Africa | 1 | 1 | 0 | 2
  Israel | 3 | 4 | 6 | 13
  United Kingdom | 0 | 1 | 0 | 1
  Italy | 1 | 1 | 0 | 2
  Serbia | 2 | 2 | 2 | 6
  Mexico | 3 | 2 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Spleen Volume
Description: Spleen volume measured by MRI
Time Frame: Spleen Volume at Baseline and Months 12, 24, and 36
Population: Intent to treat. In the Switchover group, two patients did not have MRI and one patient was splenectomized.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Naive 60 Units/kg: Patients previously naive to enzyme replacement therapy treated in Study PB-06-001 with taliglucerase alfa 60 units/kg
Arm/Group | Naive 30 Units/kg | Naive 60 Units/kg | Switchover
Number analyzed (Participants) | 12 | 14 | 15
mL
  Baseline | 2324.0 (1209.0) | 2120.0 (1426.5) | 778.0 (666.3)
  Month 12 | 1707.7 (1069.5) | 1267.9 (1114.1) | 883.7 (760.0)
  Month 24 | 1420.4 (852.3) | 946.7 (699.6) | 609.1 (442.7)
  Month 36 | 1237.2 (695.7) | 761.0 (556.0) | 548.2 (433.7)

2. Secondary Outcome: Liver Volume
Description: Liver volume measured by MRI
Time Frame: Liver volume at Baseline and Months 12, 24 and 36
Population: Intent to treat. In the Switchover group, two patients did not have MRI .
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Naive 30 Units/kg | Naive 60 Units/kg | Switchover
Number analyzed (Participants) | 12 | 14 | 16
mL
  Baseline | 2999.7 (779.4) | 2470.5 (484.9) | 1775.7 (434.4)
  Month 12 | 2515.6 (642.1) | 2118.7 (318.1) | 1788.9 (378.0)
  Month 24 | 2362.8 (518.7) | 1998.2 (291.9) | 1757.1 (357.0)
  Month 36 | 2341.1 (553.4) | 1971.8 (404.7) | 1821.2 (523.6)

3. Other Pre Specified Outcome: Spleen Volume Multiples of Normal (MN)
Description: Spleen volume measured by MRI. Normal spleen volume is 2 mL/kg × body weight (kg)
Time Frame: Baseline and Months 12, 24, and 36
Population: Intent to treat. In the Switchover group, two patients did not have MRI and one patient was splenectomized.
Measure: Mean (Standard Deviation); unit: Multiples of Normal Spleen Volume
Arm/Group | Naive 30 Units/kg | Naive 60 Units/kg | Switchover
Number analyzed (Participants) | 12 | 14 | 15
Multiples of Normal Spleen Volume
  Baseline | 16.4 (8.3) | 16.8 (14.2) | 5.5 (5.4)
  Month 12 | 11.7 (7.2) | 9.3 (9.4) | 7.0 (6.8)
  Month 24 | 9.6 (1.6) | 6.6 (5.3) | 4.0 (2.7)
  Month 36 | 8.2 (4.4) | 5.6 (4.5) | 3.7 (2.9)

4. Other Pre Specified Outcome: Liver Volume Multiples of Normal (MN)
Description: Liver volume measured by MRI. Normal liver volume is 25 mL/kg × body weight (kg).
Time Frame: Baseline and Months 12, 24 and 36
Population: Intent to treat. In the Switchover group, two patients did not have MRI.
Measure: Mean (Standard Deviation); unit: Multiples of Normal Liver Volume
Arm/Group | Naive 30 Units/kg | Naive 60 Units/kg | Switchover
Number analyzed (Participants) | 12 | 14 | 16
Multiples of Normal Liver Volume
  Baseline | 1.7 (0.4) | 1.5 (0.4) | 1.0 (0.1)
  Month 12 | 1.4 (0.3) | 1.2 (0.2) | 1.1 (0.2)
  Month 24 | 1.3 (0.2) | 1.1 (0.2) | 0.9 (0.2)
  Month 36 | 1.3 (0.2) | 1.1 (0.2) | 1.0 (0.3)

5. Secondary Outcome: Hemoglobin
Time Frame: Hemoglobin at Baseline and Months 12, 24 and 36
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Naive 30 Units/kg | Naive 60 Units/kg | Switchover
Number analyzed (Participants) | 12 | 14 | 18
mg/dL
  Baseline | 12.5 (1.8) | 11.4 (2.7) | 13.6 (1.6)
  Month 12 | 14.2 (1.7) | 13.6 (2.6) | 13.6 (1.7)
  Month 24 | 13.8 (1.6) | 13.8 (1.8) | 13.5 (1.2)
  Month 36 | 14.3 (1.5) | 14.1 (2.2) | 13.3 (1.2)

6. Secondary Outcome: Platelet Count
Time Frame: Platelet count at Baseline and Months 12, 24 and 36
Measure: Mean (Standard Deviation); unit: Platelets per cubic millimeter
Arm/Group | Naive 30 Units/kg | Naive 60 Units/kg | Switchover
Number analyzed (Participants) | 12 | 14 | 18
Platelets per cubic millimeter
  Baseline | 64900 (30133) | 69043 (28242) | 163833 (88882)
  Month 12 | 80325 (41806) | 122857 (53857) | 145250 (97426)
  Month 24 | 93333 (53328) | 141071 (73896) | 174200 (100483)
  Month 36 | 94683 (47526) | 144417 (55190) | 172467 (89340)

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Naive 30 Units/kg | Naive 60 Units/kg | Switchover
Serious Adverse Events (participants affected / at risk) | 2/12 | 2/14 | 3/18
Other Adverse Events (participants affected / at risk) | 12/12 | 12/14 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naive 30 Units/kg (N=12) | Naive 60 Units/kg (N=14) | Switchover (N=18)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Surgery: Left knee arthroscopy - Not Related
AUTOIMMUNE THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Not Related
HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — pain due to hemangioma left knee - Not Related
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Head trauma - Not Related
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Right acetabular necrosis - Not Related
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Not Related
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Not Related
RENAL STONE REMOVAL (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Not Related
TONSILLECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Not Related
TOOTH EXTRACTION (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Not Related
VOCAL CORD POLYPECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Not Related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naive 30 Units/kg (N=12) | Naive 60 Units/kg (N=14) | Switchover (N=18)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 4 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
ENDODONTIC PROCEDURE (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 2 (2) | 2 (2) | 2 (2)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
HEADACHE (Nervous system disorders) | 4 (4) | 3 (3) | 2 (2)
HYPERTENSION (Vascular disorders) | 2 (2) | 3 (3) | 1 (1)
LIMB INJURY (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 3 (3) | 7 (7)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
PAIN (General disorders) | 2 (2) | 1 (1) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 2 (2)
PHARYNGITIS (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 3 (3) | 4 (4)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
SINUSITIS (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 3 (3) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No